CLINICAL TRIAL: NCT06789185
Title: Effects of Esketamine at Subanesthetic Dose on Emergence Delirium in Preschool Children Undergoing Ambulatory Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qiu jinpeng (Other)
Responsible Party: Sponsor-Investigator, Qiu jinpeng, attending anesthesiologist, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-IRB-0377-P-01
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group S1 (0.1mg/kg esketamine) (Experimental)
  Interventions: Drug: 0.1mg/kg esketamine
- group S2 (0.2mg/kg esketamine) (Experimental)
  Interventions: Drug: 0.2mg/kg esketamine
- group C (0.1ml/kg Normal saline) (Placebo Comparator)
  Interventions: Drug: 0.1ml/kg normal saline

INTERVENTIONS:
Drug: 0.1mg/kg esketamine — Intravenous injection 0.1mg/kg esketamine about 5min before the end of the surgery
  Arms: group S1 (0.1mg/kg esketamine)
Drug: 0.2mg/kg esketamine — Intravenous injection 0.2mg/kg esketamine about 5min before the end of the surgery
  Arms: group S2 (0.2mg/kg esketamine)
Drug: 0.1ml/kg normal saline — Intravenous injection 0.1ml/kg normal saline about 5min before the end of the surgery
  Arms: group C (0.1ml/kg Normal saline)

SUMMARY:
Emergence delirium (ED) is a manifestation of acute postoperative brain dysfunction that occurs with a relatively high frequency after pediatric anesthesia. The incidence varies depending on the diagnostic criteria used and the combination of administered anesthetic drugs. The goal of this clinical trial is to investigate whether a subanesthetic dose of esketamine can reduce incidence of ED.

ELIGIBILITY:
Inclusion Criteria:

1. laparoscopic inguinal hernia repair under general anesthesia
2. aged 24~71 months
3. American Society of Anesthesiologists Physical Status I or II
4. body mass index for age between the 5th and 85th percentiles

Exclusion Criteria:

1. allergy to esketamine
2. abnormal liver or kidney function
3. glaucoma or neurological disorders
4. cardiovascular or endocrine dysfunction
5. asthma or respiratory infection in the last 2 weeks
6. developmental delay

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
The incidence of emergence delirium | Within up to 30 minutes after emergence from anesthesia
  The pediatric anesthesia emergence delirium scale consists of four items. Each item is scored 0-4 yielding a total between 0 and 20. The degree of emergence delirium increased directly with the total score. Pediatric anesthesia emergence delirium scores ≥10 at any time indicates presence of emergence delirium.

SECONDARY OUTCOMES:
Tracheal catheter extubation time | Within up to 30 minutes after operation
  The time from the cessation of sevoflurane to the point when the tracheal catheter would be remove.
emergence from anesthesia time | Within up to 30 minutes after operation
  The time from the cessation of sevoflurane to the point when the child would respond to sound stimuli or open their eyes.
The incidence of postoperative pain | Within up to 30 minutes after operation
  The FLACC scale consists of five items. Each item is scored 0-2 yielding a total between 0 and 10. The degree of pain increased directly with the total score. FLACC scores 4 or greater indicates presence of emergence delirium.
Recovery time | Within up to 50 minutes after operation
  The time from the cessation of sevoflurane to the point when the child was awakened and responded readily to their name spoken in a normal tone of voice.
The incidence of adverse effects | 24 hours after surgery.
  Postoperative nausea, vomiting, salivation, bradycardia, hypotension, and respiratory depression within 24 hours after surgery.
Blood pressure | Intraoperative and up to postoperative 20 minutes
  Blood pressure of children were measured at 0min, 5min, 10min and 20min after injection of study drug or normal saline.
heart rate | Intraoperative and up to postoperative 20 minutes
  heart rate of children were measured at 0min, 5min, 10min and 20min after injection of study drug or normal saline.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China